CLINICAL TRIAL: NCT02291380
Title: A Multi-center, Randomized, Double-blind, Placebo Parallel-Controlled Clinical Study to Evaluate the Safety and Efficacy of Botulinum Toxin Type A for Injection (HengLi ®) for Prophylactic Treatment of Chronic Migraine in Adults
Brief Title: A Study to Evaluate Botulinum Toxin Type A for Injection（HengLi®）for Prophylactic Treatment of Chronic Migraine
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lanzhou Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HengLi003
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Chronic Migraine
Keywords: Chronic Migraine; Botulinum Toxin Type A for Injection
MeSH Terms: interventions — Botulinum Toxins, Type A; Injections; Hengli BTX-A

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum Toxin Type A for Injection (Active Comparator): Botulinum Toxin Type A is a specific formulation of a locally injected muscle relaxant whose active ingredient is botulinum toxin type A produced by clostridium botulinum A strain Hall. Excipients contain sucrose, dextran and gelatin.
  Interventions: Drug: Botulinum Toxin Type A for Injection
- Placebo (Placebo Comparator): The placebo does not include botulinum toxin A ,but includes sucrose, dextran and gelatin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A for Injection — In these studies ,patients received a minimum intramuscular (IM) dose of 155 U of Botulinum Toxin Type A（HengLi®）administered to 31 injection sites across 7 head and neck muscles using a fixed-site, fixed-dose injection paradigm (each injection was 5 U in 0.1 mL). In addition, up to 40 U Botulinum Toxin Type A,administered IM to 8 additional injection sites across 3 head and neck muscles, was allowed, using a follow-the-pain approach. Thus, the minimum dose was 155 U and the maximum dose was 195 U. In the core phase, two doses of HengLi® will be injected.In the extension phase, three doses of HengLi® will be injected.
  Other Names: HengLi®
  Arms: Botulinum Toxin Type A for Injection
Drug: Placebo — In these studies, patients received placebo administered to 31 injection sites across 7 head and neck muscles using a fixed-site, fixed-dose injection paradigm (each injection was 0.1 mL). In addition, up to 0.8 mL placebo, administered IM to 8 additional injection sites across 3 head and neck muscles, was allowed, using a follow-the-pain approach. In the core phase, two doses of placebo will be injected.
  Arms: Placebo

SUMMARY:
A study, multi-center, randomized, double-blind, placebo parallel-controlled method, will be carried out to evaluate the safety and efficacy of Botulinum Toxin Type A for injection (HengLi®) for prophylactic treatment with chronic migraine in adults. In the core phase, two treatments of HengLi® or the placebo will be administrated (randomized at a ratio of 2:1, the target number is 288 subjects). In the extension phase, three treatments of HengLi® will be still administrated on 288 subjects recruited ever.

DETAILED DESCRIPTION:
Subjects in the core phase will be randomized into two groups: Botulinum Toxin Type A (HengLi®) (155U to 195U) or placebo. Study include a 28-day baseline screening period, a 24-week core phase with 2 administrations, and a 32-week extension phase with 3 administrations .Subjects enrolled will get a e-headache-diary in recording their headache symptoms and acute headache medications.

HengLi® was administered as 31 fixed-site, fixed-dose (5U), i.m. injections across 7 specific head/neck muscle areas every 12 weeks (weeks 0, 12, 24, 36, and 48). At the investigator's discretion, up to 40 U of additional HengLi® could have been administered among 3 muscle groups (occipitalis, temporalis, or trapezius) using a protocol-defined paradigm. Hence the maximum dose per treatment cycle was 195 U over 39 sites.

Efficacy Outcome Measures should be evaluated by headache diary, HIT-6 score and MIDAS score . The primary Outcome Measure: Change from baseline in the average number of days with headache per month (The last 4 weeks during the core phase and the 4 weeks during the baseline period should be compared with the number of headache days per month on average.)

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 and ≤65, male or female;
* Subjects voluntarily sign the informed consent.
* Patients complying with the ICHD-3(β) diagnostic criteria for chronic migraine.

Exclusion Criteria:

* Females who are pregnant, nursing, or planning a pregnancy during the study period, or females of childbearing potential, not using a reliable means of contraception;
* Known allergy or sensitivity to study medication or its component;
* Subjects having accepted prophylactic treatments of migraine (e.g. propranolol, metoprolol, bisoprolol, flunarizine, valproate, topiramate, gabapentin, naproxen, aspirin, amitriptyline, candesartan, lisinopril, etc.) within the 4 weeks before screening;
* Subjects with cardiac functional insufficiency;
* Subjects with renal insufficiency (serum creatinine>1.5 times ULN);
* Subjects with hepatic diseases (ALT or AST>twice ULN);
* Subjects with systemic myoneural junction diseases (e.g. myasthenia, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, etc.);
* Subjects with a history of facial palsy;
* Infection or dermatological condition at the injection sites;
* Patients with other types of migraine that do not comply with the diagnostic criteria for chronic migraine;
* Subjects ever took any type of botulinum toxin therapy in the past 6 months;
* Subjects who have used aminoglycoside antibiotics in the recent week or need to use aminoglycoside antibiotics during conduct of the clinical study;
* Subjects live with severe cognitive disorder or mental illness, outcomes will not be measured objectively;
* Subjects live with alcohol or drug abuse;
* Subjects who have been involved in other clinical studies over the 3 months prior to this study;
* Investigator's opinion that the subject has a concurrent condition(s) that may put the subject at significant risk, may confound the study results, or may interfere significantly with the conduct of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in average number of days with headache per month | Baseline (week -4 to 0) and core phase (week 21 to 24)
  The last 4 weeks during the core phase and the 4 weeks during the baseline period should be compared with the number of headache days per month on average.

SECONDARY OUTCOMES:
the average number of days with headache per month | Baseline and Week 4, 8, 12, 16, 20, 28, 32, 36, 40, 44, 48, 52, 56
  Change in the average number of days with headache per month versus the baseline
the average frequency of headache per month | Baseline and Week 4,8,12,16,20,24,28,32,36,40,44,48,52,56
  Change in the average frequency of headache per month versus the baseline
the average frequency of migraine per month | Baseline and Week 4,8,12,16,20,24,28,32,36,40,44,48,52,56
  Change in the average frequency of migraine per month versus the baseline
Proportions of subjects | Baseline and Week 4,8,12,16,20,24,28,32,36,40,44,48,52,56
  Proportions of subjects with a reduction in the average frequency of migraine per month≥50% and ≥30%
Change in the average frequency of needing emergency analgesics per month | Baseline and Week 4,8,12,16,20,24,28,32,36,40,44,48,52,56
  The number of days with the need of emergency analgesics during the observation period divided by the number of days in the observation period and multiplied by 28. The need of emergency analgesics refers to use of analgesics in case of attacks or use of drugs in advance to prevent pain attacks.
Change in the average severity of migraine | Baseline and Week 4,8,12,16,20,24,28,32,36,40,44,48,52,56
  Sum of severity scores of migraine episodes during the observation period divided by the number of migraine episodes. The severity of each migraine episode is the severity when the pain is the fiercest, expressed using VAS (0-10).
Change in the average duration of migraine | Baseline and Week 4,8,12,16,20,24,28,32,36,40,44,48,52,56
  Sum of durations of migraine episodes during the observation period divided by the number of migraine episodes.
Migraine Disability Assessment Questionnaire score(MIDAS) | Week 0,12,24,36,48,56
  Change in the MIDAS per month versus the baseline
Headache Impact Test (HIT) | Week0,4,8,12,16,20,24,28,32,36,40,44,48,52,56
  Change in the HIT per month versus the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sheng yuan Yu, Study Director — The General Hospital of People's Liberation Army(301 hospital)

IPD SHARING:
Plan to Share IPD: No